CLINICAL TRIAL: NCT00313586
Title: A Randomized Phase II Trial of Azacitidine With or Without the Histone Deacetylase Inhibitor Entinostat for the Treatment of Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia (Dysplastic Type), and Acute Myeloid Leukemia With Multilineage Dysplasia
Brief Title: Azacitidine With or Without Entinostat in Treating Patients With Myelodysplastic Syndromes, Chronic Myelomonocytic Leukemia, or Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01077; NCI-2009-01077 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E1905; CDR0000466186; E1905 (Other: ECOG-ACRIN Cancer Research Group); E1905 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p22;q23); MLLT3-MLL; Adult Acute Promyelocytic Leukemia With t(15;17)(q22;q12); PML-RARA; Alkylating Agent-Related Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndrome; Previously Treated Myelodysplastic Syndrome; Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndrome; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute | interventions — Azacitidine; entinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (azacitidine) (Experimental): Patients receive azacitidine SC QD on days 1-10. Treatment repeats every 28 days for 6-24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Other: Laboratory Biomarker Analysis
- Arm B (azacitidine, entinostat) (Experimental): Patients receive azacitidine as in Arm A and entinostat PO on days 3 and 10. Treatment repeats every 28 days for 6-24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Entinostat; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Azacitidine — Given SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS-275; SNDX-275
  Arms: Arm B (azacitidine, entinostat)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies azacitidine with or without entinostat to see how well they work compared to azacitidine alone in treating patients with myelodysplastic syndromes, chronic myelomonocytic leukemia, or acute myeloid leukemia. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Entinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving azacitidine together with entinostat may work better in treating patients with myelodysplastic syndromes, chronic myelomonocytic leukemia, or acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the overall response rate (complete, partial, and hematologic improvement-major by International Working Group [IWG] criteria) in response to azacitidine and entinostat.

II. To estimate the major response rate (complete and partial responses by the IWG response criteria) to a 10-day regimen of azacitidine and to the same regimen of azacitidine in combination with entinostat administered orally on days 3 and 10 of each cycle in patients with de novo myelodysplastic syndromes (MDS), chronic myelomonocytic leukemia (CMMoL) (dysplastic) and acute myeloid leukemia with trilineage dysplasia (AML-TLD), as well as in patients with treatment-induced MDS, CMMoL (dysplastic) and AML-TLD.

SECONDARY OBJECTIVES:

I. To evaluate the toxicity of azacitidine and entinostat in this patient population.

II. To identify changes in gene promoter methylation and gene expression which may be associated with response to azacitidine and entinostat.

III. To identify other molecular mechanisms (such as deoxyribonucleic acid [DNA] damage) which may be associated with response to azacitidine and entinostat.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive azacitidine subcutaneously (SC) once daily (QD) on days 1-10.

ARM B: Patients receive azacitidine as in Arm A and entinostat orally (PO) on days 3 and 10.

In both arms, treatment repeats every 28 days for 6-24 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* The following diagnoses will be eligible for this study:
* Myelodysplastic syndromes: the diagnosis of MDS must be confirmed by a bone marrow aspirate and/or biopsy within two weeks prior to registration; NOTE: blast count must be < 20%; patients with any International Prognostic Score (IPSS) are eligible; patients with low or intermediate (INT)-1 IPSS must have a platelet count < 50,000/mm^3 and/or absolute neutrophil count (ANC) < 500/mm^3 within seven days prior to registration
* Chronic myelomonocytic leukemia (dysplastic subtype): the diagnosis of CMMoL must be confirmed by a bone marrow aspirate and/or biopsy within two weeks prior to registration; patients with CMMoL must have a WBC < 12,000/mm^3, documented within 4 weeks prior to study entry (two sets of counts that are 2 weeks apart will be taken)
* Acute myeloid leukemia with multilineage dysplasia: the diagnosis of AML-TLD must be confirmed by a bone marrow aspirate and/or biopsy within two weeks prior to registration; NOTE: there must be evidence of >= 20% blasts on the review of the bone marrow aspirate and/or biopsy; AML-TLD will be interpreted to include patients formerly diagnosed by French-American-British (FAB) criteria as refractory anemia with excess blasts in transformation (RAEB-t), as well as patients with no history of antecedent hematologic disorder who have AML which meets criteria for AML-TLD by World Health Organization (WHO) criteria; patients with AML-TLD must have a white blood cell (WBC) =< 30,000/mm^3 documented within 4 weeks prior to study entry (two sets of counts that are 2 weeks apart will be taken); patients whose WBC has doubled within this period of time and is greater than 20,000/mm^3 at the time of screening will not be eligible
* Women must not be pregnant or breast-feeding; all females of childbearing potential must have a blood test or urine study within two weeks prior to registration to rule out pregnancy
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception
* Patient must have Eastern Cooperative Oncology Group (ECOG) performance status between 0-2
* Patient must have no prior treatment with azacitidine, decitabine or entinostat
* Patients must not have active infections at the time of registration
* Serum creatinine < 2.0 mg/dL; test must be done within seven days prior to registration
* Total serum bilirubin within institutional limits unless due to intra- or extramedullary hemolysis or Gilbert's syndrome; test must be done within seven days prior to registration
* Aspartate transaminase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine transaminase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN); tests must be done within seven days prior to registration
* Patients must not have received any AML induction chemotherapy or stem cell transplantation; any other treatment for their disease, including hematopoietic growth factors may not be given, within three weeks prior to registration, and should have recovered from all toxicities of prior therapy (to grade 0 or 1)
* Patients must have no clinical evidence of central nervous system (CNS) or pulmonary leukostasis, disseminated intravascular coagulation, or CNS leukemia
* Patients must have no serious or uncontrolled medical conditions
* Patients who have therapy-induced MDS, CMMoL (dysplastic) and AML-TLD are eligible and will be treated as separate cohorts from the patients with de novo MDS, CMMoL (dysplastic) and AML-TLD
* Patients should have a life expectancy of at least six months
* Patients must not have advanced malignant hepatic tumors
* Patients must not have a known hypersensitivity to azacitidine or mannitol
* Southwest Oncology Group (SWOG) ONLY: all SWOG patients must be registered on SWOG-9007 ("Cytogenetic Studies in Leukemia Patients"); collection of the pretreatment bone marrow specimen (or of peripheral blood if the marrow is not aspirable) must be completed within 28 days before registration; the pretreatment specimen must be submitted to a SWOG-approved cytogenetics laboratory as described in protocol SWOG-9007; note that submission of bone marrow cytogenetic studies are required to calculate the IPSS score (stratification issue); in addition, cytogenetic response will be measured at follow-up requiring a second cytogenetic study at the end of protocol treatment; NOTE: In addition to SWOG-9007, SWOG patients must be offered participation in S9910, the leukemia centralized reference laboratories and tissue repositories ancillary study; If consent is given, collection of pretreatment blood and/or marrow specimens must be completed within 14 days prior to registration. If the patient consents to participate in S9910, pretreatment specimens of marrow and/or peripheral blood must be submitted to the Southwest Oncology Group Myeloid Repository at the University of New Mexico for cellular and molecular studies; S9910 also requests submission of remission and relapse specimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2006-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Gore, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (234):
- United States (234):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Los Angeles Oncology Institute, Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Rush - Copley Medical Center, Aurora, Illinois
  - MacNeal Hospital and Cancer Center, Berwyn, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Presence Saint Joseph Hospital-Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Edward H Kaplan MD and Associates, Skokie, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Shawnee Mission Medical Center-KCCC, Shawnee Mission, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Veterans Administration, Columbia, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Ocean Medical Center, Brick, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Adirondack Cancer Center, Glens Falls, New York
  - Northwell Health NCORP, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Orange Regional Medical Center, Middletown, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Zale Lipshy University Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Medical Consultants Limited, Milwaukee, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Prebet T, Sun Z, Ketterling RP, Zeidan A, Greenberg P, Herman J, Juckett M, Smith MR, Malick L, Paietta E, Czader M, Figueroa M, Gabrilove J, Erba HP, Tallman MS, Litzow M, Gore SD; Eastern Cooperative Oncology Group and North American Leukemia intergroup. Azacitidine with or without Entinostat for the treatment of therapy-related myeloid neoplasm: further results of the E1905 North American Leukemia Intergroup study. Br J Haematol. 2016 Feb;172(3):384-91. doi: 10.1111/bjh.13832. Epub 2015 Nov 18. PMID 26577691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG member institutions between August 18, 2006 and April 29, 2011. One hundred and fifty non-treatment-induced patients and forty-seven treatment-induced patients were enrolled.
Groups:
- Arm A (Azacitidine; Non-treatment-induced Cohort): Non-treatment-induced patients receive azacitidine (50 mg/m2) subcutaneously once daily on days 1-10 in a 28-day cycle.
- Arm B (Azacitidine + Entinostat; Non-treatment-induced Cohort): Non-treatment-induced patients receive azacitidine as in arm A and oral entinostat (4 mg/m2) on days 3 and 10 of each 28-day cycle.
- Arm A (Azacitidine; Treatment-induced Cohort): Treatment-induced patients receive azacitidine (50 mg/m2) subcutaneously once daily on days 1-10 in a 28-day cycle.
- Arm B (Azacitidine + Entinostat; Treatment-induced Cohort): Treatment-induced patients receive azacitidine as in arm A and oral entinostat (4 mg/m2) on days 3 and 10 of each 28-day cycle.
Period: Overall Study
Arm/Group | Arm A (Azacitidine; Non-treatment-induced Cohort) | Arm B (Azacitidine + Entinostat; Non-treatment-induced Cohort) | Arm A (Azacitidine; Treatment-induced Cohort) | Arm B (Azacitidine + Entinostat; Treatment-induced Cohort)
Started | 75 | 75 | 24 | 23
Treated | 74 | 75 | 24 | 23
Completed | 5 | 5 | 0 | 0
Not Completed | 70 | 70 | 24 | 23
Not completed — Disease progression | 14 | 19 | 10 | 3
Not completed — Adverse Event | 12 | 18 | 3 | 10
Not completed — Death | 11 | 8 | 1 | 7
Not completed — Withdrawal by Subject | 13 | 6 | 6 | 2
Not completed — Alternative therapy | 3 | 6 | 2 | 0
Not completed — Other complicating disease | 2 | 2 | 0 | 0
Not completed — Did not achieve HI-major/better response | 10 | 7 | 2 | 1
Not completed — Physician Decision | 2 | 1 | 0 | 0
Not completed — Absolute neutrophil count not recovered | 2 | 1 | 0 | 0
Not completed — Lost insurance | 0 | 1 | 0 | 0
Not completed — Moved | 0 | 1 | 0 | 0
Not completed — Death before starting treatment | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated patients were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Azacitidine; Non-treatment-induced Cohort) | Arm B (Azacitidine + Entinostat; Non-treatment-induced Cohort) | Arm A (Azacitidine; Treatment-induced Cohort) | Arm B (Azacitidine + Entinostat; Treatment-induced Cohort) | Total
Number analyzed (Participants) | 74 | 75 | 24 | 23 | 196
Age, Continuous [Median (Full Range); unit: years] | 72 [25 to 87] | 72 [30 to 86] | 68 [54 to 83] | 71 [39 to 81] | 71 [25 to 87]
Gender [Count of Participants; unit: Participants]
  Female | 24 | 23 | 15 | 11 | 73
  Male | 50 | 52 | 9 | 12 | 123
Region of Enrollment [Number; unit: participants]
  United States | 74 | 75 | 24 | 23 | 196

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Clinical Response
Description: Clinical response is defined as a complete response (CR), partial response (PR) or trilineage response (TR) graded according to the following criteria:
  1. World Health Organization classification of the acute leukemias and myelodysplastic syndrome (by Bennett)
  2. Myelodysplastic syndromes standardized response criteria: further definition (by Cheson et al.)
  3. Report of an international working group to standardize response criteria for myelodysplastic syndromes (by Cheson et al.)
Time Frame: Assessed every 3 months if patient is < 2 years from study entry, every 6 months if patient is 2 - 5 years from study entry.
Population: All treated patients are included in the analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm A (Azacitidine; Non-treatment-induced Cohort) | Arm B (Azacitidine + Entinostat; Non-treatment-induced Cohort) | Arm A (Azacitidine; Treatment-induced Cohort) | Arm B (Azacitidine + Entinostat; Treatment-induced Cohort)
Number analyzed (Participants) | 74 | 75 | 24 | 23
Proportion of patients | 0.32 [0.22 to 0.44] | 0.27 [0.17 to 0.39] | 0.46 [0.26 to 0.67] | 0.17 [0.05 to 0.39]

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Groups:
- Arm A (Azacitidine): Patients receive azacitidine (50 mg/m2) subcutaneously once daily on days 1-10 in a 28-day cycle.
- Arm B (Azacitidine + Entinostat): Patients receive azacitidine as in arm A and oral entinostat (4 mg/m2) on days 3 and 10 of each 28-day cycle.
Arm/Group | Arm A (Azacitidine) | Arm B (Azacitidine + Entinostat)
Serious Adverse Events (participants affected / at risk) | 92/99 | 93/98
Other Adverse Events (participants affected / at risk) | 96/99 | 97/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Azacitidine) (N=99) | Arm B (Azacitidine + Entinostat) (N=98)
Autoimmune reaction (Immune system disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 55 | 54
Hemolysis (Blood and lymphatic system disorders) | 0 | 1
Leukocytes (Investigations) | 69 | 65
Lymphopenia (Investigations) | 5 | 7
Neutrophils (Investigations) | 78 | 72
Platelets (Investigations) | 75 | 76
Heart block 3rd degree (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2
Hypotension (Vascular disorders) | 4 | 3
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 | 1
Pericardial effusion (non-malignant) (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 10 | 21
Weight loss (Investigations) | 0 | 1
Constitutional, other (General disorders) | 0 | 1
DIC (Blood and lymphatic system disorders) | 1 | 0
Coagulation-other (Investigations) | 0 | 1
Injection site reaction (General disorders) | 2 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Death - multiorgan failure (General disorders) | 1 | 1
Death - sudden death (General disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 4
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 4 | 3
Ileus (Gastrointestinal disorders) | 0 | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 2 | 0
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 5
Obstruction, small bowel NOS (Gastrointestinal disorders) | 0 | 1
Typhlitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
CNS, hemorrhage (Nervous system disorders) | 0 | 1
Abdomen, hemorrhage NOS (Gastrointestinal disorders) | 0 | 1
Lower GI, hemorrhage NOS (Gastrointestinal disorders) | 0 | 1
Oral cavity, hemorrhage (Gastrointestinal disorders) | 0 | 1
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Colitis, infectious (e.g. C.diff) (Infections and infestations) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 20 | 25
Infection w/ gr3-4 neut, abdomen NOS (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, anal/perianal (Infections and infestations) | 0 | 1
Infection w/ gr3-4 neut, bronchus (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, catheter relate (Infections and infestations) | 2 | 1
Infection w/ gr3-4 neut, colon (Infections and infestations) | 0 | 1
Infection w/ gr3-4 neut, foreign body (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, lung (Infections and infestations) | 8 | 9
Infection w/ gr3-4 neut, muscle (Infections and infestations) | 0 | 1
Infection w/ gr3-4 neut, pharynx (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, sinus (Infections and infestations) | 1 | 1
Infection w/ gr3-4 neut, skin (Infections and infestations) | 1 | 2
Infection w/ gr3-4 neut, soft tissue NOS (Infections and infestations) | 0 | 1
Infection w/ gr3-4 neut, upper airway (Infections and infestations) | 1 | 1
Infection w/ gr3-4 neut, urinary tract (Infections and infestations) | 0 | 2
Infection Gr0-2 neut, catheter (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, colon (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, lung (Infections and infestations) | 1 | 2
Infection Gr0-2 neut, muscle (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, skin (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, wound (Infections and infestations) | 1 | 0
Infection w/ unk ANC abdomen NOS (Infections and infestations) | 1 | 0
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 1 | 1
Opportunistic infection lymphopenia>=gr1 (Infections and infestations) | 0 | 3
Infection w/ gr3-4 neut, blood (Infections and infestations) | 2 | 5
Infection Gr0-2 neut, blood (Infections and infestations) | 1 | 1
Infection-other (Infections and infestations) | 0 | 2
Edema limb (General disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 7
Alkaline phosphatase (Investigations) | 1 | 0
ALT, SGPT (Investigations) | 0 | 4
AST, SGOT (Investigations) | 1 | 5
Bilirubin (Investigations) | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 3
Creatinine (Investigations) | 1 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 7
Lipase (Investigations) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 12
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Neuropathy CN II vision (Eye disorders) | 0 | 1
Neuropathy-sensory (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Abdomen, pain (Gastrointestinal disorders) | 0 | 1
Cardiac/heart, pain (Cardiac disorders) | 0 | 1
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest/thoracic pain NOS (General disorders) | 0 | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Head/headache (Nervous system disorders) | 1 | 4
Joint, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 3
Visceral arterial ischemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Azacitidine) (N=99) | Arm B (Azacitidine + Entinostat) (N=98)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Hemoglobin (Blood and lymphatic system disorders) | 80 | 74
Leukocytes (Investigations) | 67 | 57
Lymphopenia (Investigations) | 11 | 8
Neutrophils (Investigations) | 56 | 49
Platelets (Investigations) | 63 | 57
Hypotension (Vascular disorders) | 2 | 8
Fatigue (General disorders) | 71 | 71
Fever w/o neutropenia (General disorders) | 10 | 7
Insomnia (Psychiatric disorders) | 8 | 10
Rigors/chills (General disorders) | 4 | 5
Sweating (Skin and subcutaneous tissue disorders) | 6 | 6
Weight loss (Investigations) | 8 | 15
Bruising (Injury, poisoning and procedural complications) | 6 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 9
Injection site reaction (General disorders) | 41 | 42
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5 | 7
Rash/desquamation (Skin and subcutaneous tissue disorders) | 11 | 13
Anorexia (Metabolism and nutrition disorders) | 27 | 49
Constipation (Gastrointestinal disorders) | 37 | 39
Dehydration (Metabolism and nutrition disorders) | 3 | 9
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 28 | 40
Dyspepsia (Gastrointestinal disorders) | 7 | 10
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 4 | 5
Nausea (Gastrointestinal disorders) | 49 | 55
Taste disturbance (Nervous system disorders) | 9 | 18
Vomiting (Gastrointestinal disorders) | 22 | 30
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 12
Petechiae (Skin and subcutaneous tissue disorders) | 4 | 9
Edema limb (General disorders) | 7 | 23
Hypoalbuminemia (Metabolism and nutrition disorders) | 22 | 41
Alkaline phosphatase (Investigations) | 11 | 17
ALT, SGPT (Investigations) | 15 | 12
AST, SGOT (Investigations) | 14 | 11
Bilirubin (Investigations) | 11 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 16 | 42
Creatinine (Investigations) | 18 | 26
Hyperglycemia (Metabolism and nutrition disorders) | 30 | 40
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 8
Hypokalemia (Metabolism and nutrition disorders) | 7 | 14
Hyponatremia (Metabolism and nutrition disorders) | 24 | 36
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1 | 7
Dizziness (Nervous system disorders) | 3 | 11
Neuropathy-sensory (Nervous system disorders) | 2 | 8
Abdomen, pain (Gastrointestinal disorders) | 9 | 13
Head/headache (Nervous system disorders) | 9 | 16
Joint, pain (Musculoskeletal and connective tissue disorders) | 3 | 10
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less